CLINICAL TRIAL: NCT00082212
Title: A Phase II Trial of Single-agent Cetuximab Dose Escalated to Rash in Patients With Persistent or Recurrent Epithelial Ovarian or Primary Peritoneal Carcinoma
Brief Title: A Study in Patients With Persistent or Recurrent Epithelial Ovarian or Primary Peritoneal Carcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to lack of sufficient efficacy.
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Chief Medical Officer, ImClone LLC
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA225-046
Record Dates: First submitted 2004-05-03; First posted 2004-05-05 (Estimated); Last update posted 2010-04-09 (Estimated); Status verified 2010-04

CONDITIONS: Ovarian Cancer
Keywords: ovarian; primary peritoneal cancer; Persistent or Recurrent Ovarian Cancer; Primary Peritoneal Carcinoma
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): 400 mg/m2 loading dose, 250 mg/m2 weekly X 2 Cycles
  Interventions: Biological: Cetuximab

INTERVENTIONS:
Biological: Cetuximab — 400 mg/m2 loading dose, 250 mg/m2 weekly X 2 Cycles
  Other Names: Erbitux

SUMMARY:
The purpose of this study is to determine the overall response rate, time to progression, and 1 yr survival with cetuximab in patients with ovarian or primary peritoneal carcinoma.

DETAILED DESCRIPTION:
To determine the overall response rate of cetuximab alone in subjects with ovarian or primary peritoneal carcinoma who have persistent or recurrent disease following 1-2 previous regimens of chemotherapy. Potential relationship between response, dose, and the occurence of rash in the treatment of subjects who have stable disease after the initial 6 weeks of treatment, time to progression, and 1 yr survival.

ELIGIBILITY:
Inclusion Criteria:

* subjects must have recurrent or persistent epithelial ovarian or primary peritoneal carcinoma. Histologic confirmation of the original primary tumor is required.
* EGFR expression must be positive as determined by an outside reference lab
* Subjects must have had a treatment-free interval following platinum of <12 mos
* All subjects must have measurable disease at baseline
* Subjects must have at least one recurrent lesion to be used to assess response
* Recovery from effect of recent surgery, radiotherapy or chemotherapy

Exclusion Criteria:

* Subjects with other invasive malignancies (including peritoneal mesotheliomas)
* Subjects with unstable cardiac disease or MI within 6 mos
* Subjects with Acute hepatitis
* Subjects with active or uncontrolled infection
* A history of prior cetuximab or other therapy which targets the EGFR pathway or prior history of prior chimerized or murine monoclonal antibody therapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2004-11; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Overall response rate | Every six weeks

SECONDARY OUTCOMES:
Relationship between response, dose, and occurence of rash | Every six weeks

CONTACTS AND LOCATIONS:
Overall Officials: E-mail: ClinicalTrials@ ImClone.com, Study Chair — Eli Lilly and Company
Locations (5):
- United States (5):
  - ImClone Investigational Site, Birmingham, Alabama
  - ImClone Investigational Site, Orlando, Florida
  - ImClone Investigational Site, New York, New York
  - ImClone Investigational Site, Philadelphia, Pennsylvania
  - ImClone Investigational Site, Seattle, Washington